CLINICAL TRIAL: NCT05182060
Title: Making Health Care Safer for Older Adults Receiving Skilled Home Health Care Services After Hospital Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00236941; 1R01HS026599-01 (AHRQ); 3R01HS026599-02S1 (AHRQ)
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Transitional Care; Frail Elderly; Home Health Care
Keywords: Transitional Care; Home Health Care; Frail Elderly; Stakeholder Participation; Quality Improvement; Medication Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transition Intervention (Experimental): We will implement a bundle of care transition safety resources with the assistance of home health coordinators at the study site.
  These resources include a link to a video about home health services, a caregiver assessment, a care task role assignment sheet, and a shopping list.
  Interventions: Behavioral: Transition Intervention
- Control (No Intervention): We will select other home health provider teams that provide care to similar populations to serve as concurrent controls.
  No interventions will be administered.

INTERVENTIONS:
Behavioral: Transition Intervention — We will implement a bundle of care transition safety strategies with the assistance of home care coordinators at the study site and corresponding home health provider teams (nurses, rehabilitation therapists).
  Home care coordinators will approach patients at the study site being referred for home health and provide resources to assist them with preparing for their transition home. These resources include a link to a video about home health services, a caregiver assessment, a care task role assignment sheet, and a shopping list. The study team will contact the older adult and caregiver by telephone within 48 hours of the home visit to confirm eligibility, explain the study, obtain consent for participation, and ask them to complete the the Hospital-to-Home Health Transition Quality Index (H3TQ) over the phone. Home health providers in the home will also complete the H3TQ.
  Arms: Transition Intervention

SUMMARY:
Care transitions are the movement of a person from one healthcare setting to another. Older adults who require skilled home health care ("home health") services (e.g., home-based nursing) after hospital discharge are at high risk of experiencing early re-hospitalization. Home health agencies need strategies to ensure safe transitions, yet there is relatively little research to guide improvement efforts. The goal of the study is to develop and test tools to allow home health agencies to identify and act upon threats to older adults' safety in real time. The investigators first analyzed threats to older adult safety during hospital-to-home health transitions and refined a bundle of interventions through stakeholder engagement. This prospective pilot will implement and measure the bundle of interventions.

DETAILED DESCRIPTION:
Using a participatory ergonomics process, the investigators will pilot a bundle of interventions developed by stakeholders in a prospective cohort study to test feasibility. The study settings and inclusion criteria will be the same as used in the investigators' initial trial: cohort study of older adults (aged ≥ 65 years) experiencing a hospital-to-home health transition to the study sites, regardless of diagnosis. The investigators will implement the bundle with the assistance of home health provider teams at the study sites. The investigators will select other home health provider teams that provide care to similar populations to serve as concurrent controls. To provide historical control data, the investigators will also collect data on patient outcomes for the past year prior to the implementation of the bundle. Intervention refinement teams (IRTs) will meet to assess the impact of the bundle.

The investigators will retrospectively extract the dependent variables going back one year before implementation of the bundle (baseline) up until one year after implementation for both intervention and control groups. Outcome measures will include 30-day emergency department (ED) visit use or re-hospitalization, and mortality. The investigators will collect independent variables (Hospital-to-Home Health Transition Quality Index (H3TQ)) and measures of bundle impact from the intervention group. The investigators developed measures of bundle impact after a review of related existing measures. The investigators will collect measures of bundle impact in two ways: (1) through online surveys sent to all home health providers and older adults involved in the bundle at the end of the study period (30 days) using a Likert-type response scale; and (2) focus groups of home health providers and older adults.

The investigators will conduct two focus groups at the study site of: (1) the home health providers implementing the bundle (approximately 5 at each site, 10 total), and (2) a subset of the older adults/caregivers receiving the bundle. The investigators will randomly select approximately 10 older adults/caregivers at each site (20 total) and call these older adults/caregivers for an invitation to participate. Focus groups will discuss on key outcomes important in implementation research, which are distinct from system and clinical treatment outcomes and serve as indicators of implementation success: (1) acceptability, (2) appropriateness, (3) identification of barriers to implementation, and (4) analysis of impact on workflow. Focus groups will last 1.5 hours and will be audio-taped and transcribed. At least two researchers will independently review each focus group transcript and identify themes and sub-themes related to each of the four measures of bundle impact.

The investigators will compare dependent variables as follows: (1) pre-post comparison of dependent variables with historical controls for intervention and control groups separately; and (2) concurrent comparison of dependent variables between intervention and control groups.

For this feasibility study, the investigators anticipate having approximately 100 patients in the intervention group over the one-year pilot period.

ELIGIBILITY:
Inclusion Criteria:

Older Adults

* Aged ≥ 65 years
* Can speak English or Spanish
* Is capable of assent
* Hospitalized on a medical or surgical service
* Referred for skilled home healthcare services (home health) after hospital discharge or skilled nursing facility (SNF) discharge

Family Caregivers

* Unpaid
* Assist the older adult with at least one healthcare task. Healthcare tasks include the following activities: managing health care bills, scheduling medical appointments, getting to and from medical appointments, getting medical equipment, getting services, getting information, following a diet, obtaining medication, planning a medication schedule, taking medication, and deciding to stop or change medication.

Home Health Providers

* Employed by participating sites
* Directly provide care to, or arrange services for, an eligible older adult

Exclusion Criteria:

* Community referrals to home health: Older adults referred to home health from the ambulatory setting (e.g., outpatient clinic) and without a recent hospitalization or SNF stay.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 761 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
ED visit use or re-hospitalization | Within 30 days after hospital discharge
  Whether or not the older adult experiences an ED visit use or re-hospitalization within 30 days of hospital discharge. This is a composite endpoint.

SECONDARY OUTCOMES:
Mortality within 30 days of hospital discharge | Within 30 days after hospital discharge
  Whether or not the older adult passes away within 30-days of hospital discharge.
Existence of Unresolved Medication Issues | Within 30 days after hospital discharge
  Existence of any medication issues (incorrect medication list, incorrect prescription, unfilled prescription, etc.) within 30 days of hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Arbaje, MD, MPH, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Division of Geriatric Medicine and Gerontology, Johns Hopkins University School of Medicine, Baltimore, Maryland, United States